CLINICAL TRIAL: NCT01459146
Title: The Impact of Intermittent Preventive Malaria Treatment With Artemisinin Combination Therapy (ACT) on Hemoglobin, Malaria, Schistosomiasis, and School Attention Among Primary Schoolchildren in the Kassena-Nankana Districts, Ghana
Brief Title: Artemisinin-based Combination Therapy-Intermittent Preventive Treatment (ACT-IPT) Trial Among Schoolchildren in Kassena-Nankana, Ghana
Acronym: ACTIPT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Navrongo Health Research Centre, Ghana (Other)
Collaborators: DBL -Institute for Health Research and Development (Other)
Responsible Party: Principal Investigator, Dr. Ernest Cudjoe Opoku M.D., M.P.H., M.D., M.P.H., Navrongo Health Research Centre, Ghana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NHRCIRB098
Record Dates: First submitted 2011-10-17; First posted 2011-10-25 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Malaria; Schistosomiasis; Helminthiasis; Anemia; Change in Sustained Attention
Keywords: IPT; malaria; ACT; schistosomiasis; Hemoglobin; Anemia; Sustained attention; Recall; Schoolchildren; Kassena-Nankana
MeSH Terms: conditions — Malaria; Schistosomiasis; Helminthiasis; Anemia | interventions — Artemether, Lumefantrine Drug Combination; Albendazole; Praziquantel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AL plus ABZ; Arm 1 (Experimental): Artemether-Lumefantrine combination 20mg/120mg 12 hourly for 3 days oral, plus albendazole 400mg stat oral
  Interventions: Drug: Artemether-lumefantrine combination plus albendazole
- AL plus PZQ plus ABZ; Arm 2 (Active Comparator): artemether-lumefantrine combination 120mg/20mg 12 hourly for 3 days; plus praziquantel 40mg/kg stat; plus albendazole 400mg stat oral
  Interventions: Drug: Artemether-lumefantrine plus Praziquantel plus Albendazole
- ABZ plus PZQ; Arm 3 (Active Comparator): Albendazole 400mg stat plus Praziquantel 40mg/kg stat oral
  Interventions: Drug: Albendazole plus Praziquantel

INTERVENTIONS:
Drug: Artemether-lumefantrine combination plus albendazole — AL: 20mg/120mg 12-hourly orally for 3 days ABZ: 400mg oral stat
  Arms: AL plus ABZ; Arm 1
Drug: Artemether-lumefantrine plus Praziquantel plus Albendazole — Artemether-lumefantrine 20mg/120mg 12 hourly for 3 days, plus praziquantel 40mg/kg stat, plus albendazole 400mg stat oral
  Arms: AL plus PZQ plus ABZ; Arm 2
Drug: Albendazole plus Praziquantel — Albendazole 400mg stat plus Praziquantel 40mg/kg stat oral
  Arms: ABZ plus PZQ; Arm 3

SUMMARY:
The purpose of this study is to determine if Artemisinin-based Combination Therapy, ACT,(artemether-lumefantrine) used as intermittent preventive treatment (IPT) alone or in combination with praziquantel, will have any effects on anemia, malaria, schistosomiasis and school sustained attention and concentration.

DETAILED DESCRIPTION:
Introduction: Malaria, schistosomiasis and soil-transmitted helminth (STH) infections are rife in sub-Saharan Africa where school children are at great risk of morbidity. Although the strategy of using intermittent preventive treatment (IPT) for malaria control has been proven beneficial among infants and pregnant women, it is yet to be implemented in school children on a large scale. Sulfadoxine-pyrimethamine (SP) use as IPT is being limited by widespread reports of resistance. Artemisinin-based combination therapy (ACT) has been proven efficacious as IPT among school children in few studies. Other studies have shown that artemisinin derivatives exhibit anti-schistosomal activity. This could be an added effect of using ACTs, as IPT, to prevent malaria related morbidity in school children in sub-Saharan Africa.

General Objective: To examine the effect of IPT with ACTs and anti-helminthes against malaria and helminthes infections on health and school attention among children 6 to 12 years old.

Specific objectives

1. To estimate the prevalence of malaria parasitemia, schistosomiasis and anemia among primary schoolchildren.
2. To determine the impact of 3 doses of IPT (with artemether-lumefantrine) and de-worming (with albendazole and/or praziquantel) on hemoglobin and school (classroom) attention and recall.
3. To determine the effects of IPT (with artemether-lumefantrine) and de-worming (with albendazole and /or praziquantel) on the prevalence and intensity of schistosomes infection among schoolchildren.
4. To determine the safety and tolerability of IPT with artemether-lumefantrine combined with albendazole and/or praziquantel among school children.

Materials and methods: An open-labeled randomized trial, including 3 arms, will be carried out in 6 primary schools in the Kassena-Nankana Districts, Ghana, where malaria and schistosome infection (with S. hematobium and S. mansoni) are endemic. After informed consent and assent are obtained, about 345 (115 in each arm) class three school children will be investigated for malaria parasitemia, anemia, schistosome and soil-transmitted helminths infections, and classroom attention and recall in a baseline pre-intervention survey. Mass treatment is then carried out in the 6 randomized schools with ACT and albendazole in one study arm; ACT, albendazole and praziquantel in the second arm while albendazole and praziquantel will be given in the third school arm. ACT mass treatment using artemether-lumefantrine is carried out every school term (4 monthly) for one year while praziquantel is given once and albendazole twice a year. After one academic year, the same 345 (115 in each arm) selected participants in class three are assessed for hemoglobin, malaria parasitemia, STH and schistosome infections and classroom attention and recall. Safety and tolerability of the combined IPT is assessed at 28 days post treatment.

Data analysis- Data will be analyzed by both intention-to-treat and per-protocol employing uni-variate and multivariate logistic regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Parental informed consent and assent by schoolchildren
* No known history of allergy to any study drug
* Aged 6 or more years

Exclusion Criteria:

* lack of parental informed consent and assent by schoolchildren
* Known allergy or history of allergy to any study drug
* Aged less than 6 years

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 345 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-10 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Prevalence and density of malaria parasites, determined by microscopy, as a measure of efficacy | Day 28 post intervention
  Change from baseline of prevalence and density of malaria parasitemia 28 days post interventions

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Day 365
  Number of reported adverse events within twelve months of intervention per study arm
Number of schoolchildren with sustained attention and recall as a measure of efficacy | Day 365
  Change in sustained classroom attention and recall in 365 days of start of intervention from baseline
Proportion of schoolchildren with anemia as a measure of safety and tolerability | Day 365
  Proportion of schoolchildren having hemoglobin level less than 12.0g/dl from baseline level in 365 days of start of intervention
Prevalence and intensity of urinary schistosomiasis as a measure of efficacy | 365 days post first intervention
  Proportion of schoolchildren with urinary schistosomiasis by study arm compared to baseline
Prevalence and density of malaria parasites by microscopy as a measure of efficacy | 365 days
  Proportion of schoolchildren with malaria parasitemia by study arm compared to baseline
Prevalence and intensity of intestinal schistosomiasis among schoolchildren as a measure of efficacy | 365 days
  Proportion of schoolchildren with intestinal schistosomiasis by study arm compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ernest C Opoku, MD, MPH, Principal Investigator — Navrongo Health Research Centre, Ghana; Pascal Magnussen, MD, Principal Investigator — University of Copenhagen; Abraham V Hodgson, MD, MPH, PhD, Study Director — Navrongo Health Research Centre, Ghana; Edmund L Browne, MD, MPH, PhD, Principal Investigator — University of Development Studies; Annette Olsen, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- NHRC, Navrongo, Ghana